CLINICAL TRIAL: NCT04338022
Title: A Phase III, Multicenter, Randomized, Parallel Group, Double Blind, Double Dummy, Active Controlled Study of Evobrutinib Compared With Teriflunomide, in Participants With Relapsing Multiple Sclerosis to Evaluate Efficacy and Safety (evolutionRMS 1)
Brief Title: Study of Evobrutinib in Participants With RMS (evolutionRMS 1)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary analysis of the RMS phase 3 study (MS200527_0080) resulted in the early termination of the study.
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS200527_0080; 2019-004972-20 (EudraCT Number)
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Evobrutinib; Teriflunomide; Aubagio®; Relapsing Multiple Sclerosis
MeSH Terms: interventions — teriflunomide; evobrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teriflunomide (Active Comparator)
  Interventions: Drug: Teriflunomide
- Evobrutinib (Experimental)
  Interventions: Drug: Evobrutinib

INTERVENTIONS:
Drug: Teriflunomide — Participants received Teriflunomide at a dose of 14 milligrams (mg) orally once daily up to 156 weeks in Double blind treatment period (DBTP) followed by once daily oral doses of Teriflunomide 14 mg up to 96 weeks in double blind extension (DBE) period and followed by once daily oral doses of Teriflunomide 14 mg up to 96 weeks in open label extension (OLE) period.
  Arms: Teriflunomide
Drug: Evobrutinib — Participants received Evobrutinib at a dose of 45 mg orally twice daily up to 156 weeks in Double blind treatment period (DBTP) followed by twice daily oral doses of Evobrutinib 45 mg up to 96 weeks in double blind extension (DBE) period and followed by twice daily oral doses of Evobrutinib 45 mg up to 96 weeks in open label extension (OLE) period.
  Other Names: M2951
  Arms: Evobrutinib

SUMMARY:
The study is to evaluate the efficacy and safety of evobrutinib administered orally twice daily versus Teriflunomide (Aubagio®), administered orally once daily in participants with Relapsing Multiple Sclerosis (RMS). Participants who complete the double-blind treatment period (DBTP) and double-blind extension period (DBEP) prior to approval of a separate long-term follow-up study in their country will get an option for evobrutinib treatment continuation through a 96-week open-label extension (OLE) period.

ELIGIBILITY:
Inclusion Criteria:

* Participants are diagnosed with RMS (relapsing-remitting multiple sclerosis [RRMS] or secondary progressive multiple sclerosis [SPMS] with relapses) in accordance with 2017 Revised McDonald criteria (Thompson 2018)
* Participants with one or more documented relapses within the 2 years before Screening with either: a. one relapse which occurred within the last year prior to randomization, OR b. the presence of at least 1 gadolinium-enhancing (Gd+) T1 lesion within 6 months prior to randomization
* Participants have Expanded Disability Status Scale (EDSS) score of 0 to 5.5 at Screening and Baseline (Day 1). Participants with an EDSS score <= 2 at Screening and Baseline (Day 1) are only eligible for participation if their disease duration (time since onset of symptoms) is no more than 10 years
* Participants are neurologically stable for >= 30 days prior to both screening and baseline (Day 1)
* Female participants must be neither pregnant nor breast-feeding or must lack child-bearing potential (as defined by either: post-menopausal or surgically sterile), or use an effective method of contraception for the duration of the study and at least 2 years after study intervention due to the long elimination period for teriflunomide of 2 years, unless the participant undergoes an accelerated elimination procedure
* Male participants must refrain from donating sperm and/or abstain from intercourse with women of child-bearing potential or use an effective method of contraception for the duration of the study and at least 2 years after study intervention due to the long elimination period for teriflunomide of 2 years, unless the participant undergoes an accelerated elimination procedure
* Participants have given written informed consent prior to any study-related procedure
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Participants diagnosed with Progressive MS, in accordance with the 2017 Revised McDonald criteria as follows: a). Participants with Primary Progressive MS. b).

Participants with secondary progressive MS without evidence of relapse

* Disease duration more than (>) 10 years in participants with an EDSS =< 2.0 at screening and Baseline (Day 1)
* Immunologic disorder other than MS, or any other condition requiring oral, intravenous (IV) , intramuscular, or intra-articular corticosteroid therapy, with the exception of well-controlled Type 2 diabetes mellitus or well controlled thyroid disease
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1124 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (279):
- United States (51):
  - Research Site 629, Mobile, Alabama
  - Research Site 614, Phoenix, Arizona
  - Research Site 677, Phoenix, Arizona
  - Research Site 642, Long Beach, California
  - Research Site 644, Pasadena, California
  - Research Site 672, San Diego, California
  - Research Site 634, Stamford, Connecticut
  - Research Site 656, Washington D.C., District of Columbia
  - Research Site 616, Boca Raton, Florida
  - Research Site 625, Maitland, Florida
  - Research Site 617, Miami, Florida
  - Research Site 643, Ormond Beach, Florida
  - Research site 645, St. Petersburg, Florida
  - Research Site 652, Tallahassee, Florida
  - Research Site 621, Elk Grove Village, Illinois
  - Research Site 649, Northbrook, Illinois
  - Research Site 675, Peoria, Illinois
  - Research Site 628, Rolling Meadows, Illinois
  - Research Site 624, Indianapolis, Indiana
  - Research Site 632, Kansas City, Kansas
  - Research Site 653, New Orleans, Louisiana
  - Research Site 623, Baltimore, Maryland
  - Research Site 633, Boston, Massachusetts
  - Research Site 639, Foxborough, Massachusetts
  - Research Site 635, Lawrence, Massachusetts
  - Research Site 636, Worcester, Massachusetts
  - Research Site 613, Detroit, Michigan
  - Research Site 612, Farmington Hills, Michigan
  - Research Site 638, St Louis, Missouri
  - Research Site 664, St Louis, Missouri
  - Research Site 668, Omaha, Nebraska
  - Research Site 626, Las Vegas, Nevada
  - Research Site 667, Audubon, New Jersey
  - Research Site 620, Patchogue, New York
  - Research Site 663, Akron, Ohio
  - Research Site 630, Toledo, Ohio
  - Research Site 611, Oklahoma City, Oklahoma
  - Research Site 641, Oklahoma City, Oklahoma
  - Research Site 615, Springfield, Oregon
  - Research Site 647, Willow Grove, Pennsylvania
  - Research Site 648, Knoxville, Tennessee
  - Research Site 627, Nashville, Tennessee
  - Research Site 637, Nashville, Tennessee
  - Research Site 662, Dallas, Texas
  - Research Site 631, Houston, Texas
  - Research Site 650, Lubbock, Texas
  - Research Site 619, Round Rock, Texas
  - Research Site 676, Layton, Utah
  - Research Site 673, Alexandria, Virginia
  - Research Site 654, Virginia Beach, Virginia
  - Research Site 651, Milwaukee, Wisconsin
- Argentina (15):
  - Research Site 561, Buenos Aires
  - Research Site 562, Buenos Aires
  - Research Site 577, Buenos Aires
  - Research Site 566, Ciudad Autonoma Buenos Aires
  - Research Site 567, Ciudad Autonoma Buenos Aires
  - Research Site 574, Ciudad Autonoma Buenos Aires
  - Research Site 579, Ciudad Autonoma Buenos Aires
  - Research Site 564, Córdoba
  - Research Site 568, Godoy Cruz
  - Research Site 565, Rosario
  - Research Site 569, Rosario
  - Research Site 571, Salta
  - Research Site 572, San Juan
  - Research Site 563, San Miguel de Tucumán
  - Research Site 576, Villa Nueva
- Australia (6):
  - Research Site 104, Auchenflower
  - Research Site 107, Concord
  - Research Site 109, Hobart
  - Research Site 101, Liverpool
  - Research Site 102, New Lambton Heights
  - Research Site 103, St Leonards
- Austria (4):
  - Research Site 151, Innsbruck
  - Research Site 156, Linz
  - Research Site 154, Salzburg
  - Research Site 153, Vienna
- Belgium (7):
  - Research Site 474, Brussels
  - Research Site 475, Brussels
  - Research Site 473, Kortrijk
  - Research Site 471, La Louvière
  - Research Site 472, Liège
  - Research Site 478, Overpelt
  - Research Site 476, Roeselare
- Bosnia and Herzegovina (3):
  - Research Site 161, Bihać
  - Research Site 163, Mostar
  - Research Site 162, Sarajevo
- Bulgaria (10):
  - Research Site 171, Pleven
  - Research Site 174, Pleven
  - Reasearch Site 175, Plovdiv
  - Research Site 177, Plovdiv
  - Research Site 172, Sofia
  - Research Site 173, Sofia
  - Research Site 176, Sofia
  - Research Site 178, Sofia
  - Research Site 179, Sofia
  - Research Site 180, Sofia
- Canada (5):
  - Research Site 126, Greenfield Park
  - Research Site 125, Lévis
  - Research Site 128, Moncton
  - Research Site 129, Montreal
  - Research Site 124, Toronto
- Colombia (4):
  - Research Site 591, Barranquilla
  - Research Site 597, Barranquilla
  - Research Site 592, Medellín
  - Research Site 600, Medellín
- Croatia (5):
  - Research Site 193, Osijek
  - Research Site 197, Rijeka
  - Research Site 195, Varaždin
  - Research Site 192, Zagreb
  - Research Site 194, Zagreb
- Czechia (12):
  - Research Site 212, Brno
  - Research Site 218, Brno
  - Research Site 219, Hradec Králové
  - Research Site 222, Hradec Králové
  - Research Site 211, Jihlava
  - Research Site 223, Ostrava
  - Research Site 215, Pardubice
  - Research Site 216, Plzen-Bory
  - Research Site 217, Prague
  - Research Site 220, Prague
  - Research Site 224, Prague
  - Research Site 213, Praha 4 - Krc
- Estonia (2):
  - Research Site 231, Tallinn
  - Research Site 232, Tartu
- Research Site 491, Turku, Finland
- France (11):
  - Research Site 510, Bron
  - Research Site 509, Caen
  - Research Site 502, Grenoble
  - Research Site 504, Lille
  - Research Site 508, Lille
  - Reserach Site 505, Montpellier
  - Research Site 511, Nantes
  - Research Site 506, Nice
  - Research Site 507, Rennes
  - Research Site 501, Rouen
  - Research Site 503, Toulouse
- Georgia (10):
  - Research Site 241, Tbilisi
  - Research Site 242, Tbilisi
  - Research Site 243, Tbilisi
  - Research Site 244, Tbilisi
  - Research Site 245, Tbilisi
  - Research Site 246, Tbilisi
  - Research Site 247, Tbilisi
  - Research Site 248, Tbilisi
  - Research Site 249, Tbilisi
  - Research Site 250, Tbilisi
- Germany (15):
  - Research Site 265, Bamberg
  - Research Site 267, Bayreuth
  - Research Site 271, Berlin
  - Research Site 264, Bochum
  - Research Site 274, Bonn
  - Research Site 270, Erbach im Odenwald
  - Research Site 268, Essen
  - Research Site 263, Frankfurt
  - Research Site 275, Hanover
  - Research Site 272, Mannheim
  - Research Site 262, München
  - Research Site 266, Münster
  - Research Site 261, Potsdam
  - Research Site 273, Siegen
  - Research Site 269, Ulm
- Hong Kong (3):
  - Research Site 700, Hong Kong
  - Research Site 704, Hong Kong
  - Research Site 701, Shatin
- Hungary (9):
  - Research Site 282, Budapest
  - Research Site 285, Budapest
  - Research Site 286, Budapest
  - Research Site 288, Budapest
  - Research Site 290, Budapest
  - Research Site 281, Kistarcsa
  - Research Site 284, Pécs
  - Research Site 289, Tatabánya
  - Research Site 291, Vác
- India (3):
  - Research Site 457, Hyderabad
  - Research Site 456, Nashik
  - Research Site 451, New Delhi
- Israel (6):
  - Research Site 303, Ashkelon
  - Research Site 305, Jerusalem
  - Research Site 307, Petah Tikva
  - Research Site 308, Ramat Gan
  - Research Site 301, Rehovot
  - Research Site 304, Safed
- Italy (12):
  - Research Site 319, Bologna
  - Research Site 321, Chieti
  - Research Site 322, Genova
  - Research Site 320, Messina
  - Research Site 315, Milan
  - Research Site 314, Montichiari
  - Research Site 316, Napoli
  - Research Site 317, Napoli
  - Research Site 311, Reggio Calabria
  - Research Site 318, Roma
  - Research Site 312, Salerno
  - Research Site 313, Verona
- Mexico (2):
  - Research Site 133, Aguascalientes
  - Research Site 134, Culiacán
- Netherlands (4):
  - Research Site 534, Hoorn
  - Research Site 531, Nieuwegein
  - Research Site 535, Rotterdam
  - Research Site 532, Sittard-Geleen
- Poland (10):
  - Research Site 332, Bydgoszcz
  - Research Site 335, Gdansk
  - Research Site 336, Katowice
  - Research Site 340, Knurów
  - Research Site 339, Lodz
  - Research Site 337, Lublin
  - Research Site 331, Oświęcim
  - Research Site 338, Rzeszów
  - Research Site 341, Warsaw
  - Research Site 342, Warsaw
- Russia (19):
  - Research Site 365, Barnaul
  - Research Site 355, Kaluga
  - Research Site 358, Kazan'
  - Research Site 354, Kirov
  - Research Site 363, Krasnoyarsk
  - Research Site 353, Moscow
  - Research Site 359, Moscow
  - Research Site 352, Nizhny Novgorod
  - Research Site 367, Perm
  - Research Site 362, Pyatigorsk
  - Research Site 356, Saint Petersburg
  - Research Site 369, Saint Petersburg
  - Research Site 360, Saratov
  - Research Site 361, Smolensk
  - Research Site 370, Tomsk
  - Research Site 351, Ufa
  - Research Site 357, Ulyanovsk
  - Research Site 366, Yaroslavl
  - Research Site 368, Yekaterinburg
- Serbia (8):
  - Research Site 382, Belgrade
  - Research Site 383, Belgrade
  - Research Site 385, Belgrade
  - Research Site 389, Kragujevac
  - Research Site 390, Niš
  - Research Site 388, Novi Sad
  - Research Site 384, Užice
  - Research Site 381, Valjevo
- South Korea (7):
  - Research Site 462, Goyang-si
  - Research Site 461, Seoul
  - Research Site 463, Seoul
  - Research Site 464, Seoul
  - Research Site 465, Seoul
  - Research Site 466, Seoul
  - Research Site 467, Seoul
- Spain (11):
  - Research Site 406, Barcelona
  - Research Site 407, Barcelona
  - Research Site 405, Cadiz
  - Research Site 402, Donostia / San Sebastian
  - Research Site 401, Lleida
  - Research Site 403, Madrid
  - Research Site 408, Madrid
  - Research Site 409, Madrid
  - Research Site 411, Pozuelo de Alarcón
  - Research Site 410, Salt
  - Research Site 404, Seville
- Taiwan (4):
  - Research site 713, Kaohsiung City
  - Research Site 711, Taichung
  - Research site 714, Taipei
  - Research site 715, Taipei
- Ukraine (16):
  - Research Site 432, Chernivtsi
  - Research Site 425, Kharkiv
  - Research Site 429, Kharkiv
  - Research Site 430, Kharkiv
  - Research Site 435, Kharkiv
  - Research Site 436, Kharkiv
  - Research Site 437, Kharkiv
  - Research Site 422, Kropyvnytskyi
  - Research Site 438, Kyiv
  - Research Site 426, Lviv
  - Research Site 424, Odesa
  - Research Site 423, Poltava
  - Research Site 427, Sumy
  - Research Site 431, Vinnytsia
  - Research Site 421, Zaporizhzhia
  - Research Site 428, Zaporizhzhia
- United Kingdom (4):
  - Research Site 544, Exeter
  - Research Site 549, Glasgow
  - Research Site 552, Newcastle
  - Research Site 547, Swansea

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Montalban X, Vermersch P, Arnold DL, Bar-Or A, Cree BAC, Cross AH, Kubala Havrdova E, Kappos L, Stuve O, Wiendl H, Wolinsky JS, Dahlke F, Le Bolay C, Shen Loo L, Gopalakrishnan S, Hyvert Y, Javor A, Guehring H, Tenenbaum N, Tomic D; evolutionRMS investigators. Safety and efficacy of evobrutinib in relapsing multiple sclerosis (evolutionRMS1 and evolutionRMS2): two multicentre, randomised, double-blind, active-controlled, phase 3 trials. Lancet Neurol. 2024 Nov;23(11):1119-1132. doi: 10.1016/S1474-4422(24)00328-4. Epub 2024 Sep 19. PMID 39307151
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200527_0080
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were enrolled in the Open Label Extension (OLE) Period after Double Blind Treatment Period (DBTP) Week 96 and they did not enter Double Blind Extension (DBE) period.
Period: Double-blind Treatment Period: 156 Weeks
Arm/Group | Teriflunomide | Evobrutinib
Started | 564 | 560
Completed | 396 | 384
Not Completed | 168 | 176
Not completed — Adverse Event | 56 | 72
Not completed — Lost to Follow-up | 6 | 5
Not completed — Lack of Efficacy | 19 | 23
Not completed — Withdrawal by Subject | 56 | 55
Not completed — Death | 1 | 1
Not completed — Protocol Non-Compliance | 5 | 5
Not completed — Other Reason | 24 | 14
Not completed — Randomized, but not treated | 1 | 1
Period: Double-blind Extension: 96 Weeks
Arm/Group | Teriflunomide | Evobrutinib
Started | 377 | 359
Completed | 371 | 346
Not Completed | 6 | 13
Not completed — Lack of Efficacy | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other Reason | 3 | 9
Period: Open Label Extension: 96 Weeks
Arm/Group | Teriflunomide | Evobrutinib
Started | 0 | 3
Completed | 0 | 0
Not Completed | 0 | 3
Not completed — Study Termination | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriflunomide | Evobrutinib | Total
Number analyzed (Participants) | 564 | 560 | 1124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (9.5) | 37 (9.6) | 38 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 377 | 751
  Male | 190 | 183 | 373
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 60 | 63 | 123
  Ethnicity-Not Hispanic or Latino | 504 | 497 | 1001
  Race-American Indian or Alaska Native | 6 | 13 | 19
  Race-Asian | 10 | 16 | 26
  Race-Black or African American | 2 | 4 | 6
  Race-Multiple | 5 | 2 | 7
  Race-Other | 2 | 1 | 3
  Race-Unknown or Not Reported | 3 | 5 | 8
  Race-White | 536 | 519 | 1055

OUTCOME MEASURES:

1. Primary Outcome: Double Blind Treatment Period (DBTP) and Double Blind Extension (DBE) Period: Annualized Relapse Rate (ARR)
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, adverse events (AEs,) and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days).
Time Frame: From baseline to 172 weeks
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 564 | 560
relapses per year | 0.13 [0.11 to 0.15] | 0.14 [0.12 to 0.16]

2. Primary Outcome: Open Label Extension (OLE) Period: Number of Participants With Adverse Events (AEs) and Serious AEs
Description: Adverse event (AE): Any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study drug. Therefore, an AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important.
Time Frame: From OLE Baseline (DBTP Week 96) to OLE Week 52
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
Participants
  Participants with AEs | 1
  Participants with Serious AEs | 0

3. Secondary Outcome: DBTP and DBE Period: Percentage of Participants Without 12-Week Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability progression was defined as increase in EDSS of greater than or equal to [>=] 1 point from baseline EDSS score, if EDSS score at baseline is 5.0 or less and an increase of >=0.5 point, if the baseline score is 5.5. Disability progression is considered sustained for 12 weeks when the initial increase in the EDSS is confirmed at a regularly scheduled visit at least 12 weeks after the initial documentation of neurological worsening. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). Kaplan-Meier method was used to estimate the percentage of participants without 12-week CDP.
Time Frame: Week 96 and Week 156 (combined DBTP and DBE period)
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. The result reported for this outcome measure are the results from data of combined DBTP and DBE periods.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 564 | 560
percentage of participants
  Week 96 | 91.0 [88.0 to 93.3] | 91.3 [88.3 to 93.5]
  Week 156 | 86.0 [81.5 to 89.5] | 87.9 [83.5 to 91.1]

4. Secondary Outcome: DBTP and DBE Period: Percentage of Participants Without 24-Week Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability progression was defined as increase in EDSS of greater than or equal to [>=] 1 point from baseline EDSS score, if EDSS score at baseline is 5.0 or less and an increase of >=0.5 point, if the baseline score is 5.5. Disability progression is considered sustained for 24 weeks when the initial increase in the EDSS is confirmed at a regularly scheduled visit at least 24 weeks after the initial documentation of neurological worsening. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). Kaplan-Meier method was used to estimate the percentage of participants without 24-week CDP.
Time Frame: Week 96 and Week 156 (combined DBTP and DBE periods)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 564 | 560
percentage of participants
  Week 96 | 94.3 [91.9 to 96.1] | 92.7 [89.9 to 94.7]
  Week 156 | 92.3 [89.2 to 94.5] | 92.1 [89.2 to 94.3]

5. Secondary Outcome: DBTP and DBE Period: Percentage of Participants With 24-Week Confirmed Disability Improvement (CDI) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability improvement was defined as a reduction of 1 point from Baseline EDSS score when the Baseline score is >= 2 and less than or equal to [<=] 6 and a reduction of 0.5 point from Baseline EDSS score when the Baseline score is >= 6.5 and <= 9.5. Disability improvement is considered sustained when the initial reduction in the EDSS score is confirmed at a regularly scheduled visit at least 24 weeks after the initial reduction. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis). Kaplan-Meier method was used to estimate the percentage of participants with 12-week CDI.
Time Frame: Week 96 and Week 156 (combined DBTP and DBE periods)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 564 | 560
percentage of participants
  Week 96 | 7.9 [5.6 to 11.2] | 9.4 [6.7 to 13.0]
  Week 156 | 8.8 [6.2 to 12.4] | 10.1 [7.3 to 13.9]

6. Secondary Outcome: DBTP and DBE Period: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Score at Week 48, Week 96, Week 120, Week 144 and Week 156
Description: Physical function was assessed with PROMISnq Short Form v2.0 - Physical Function - Multiple Sclerosis 15a (PROMISnq PF(MS) 15a). PROMISnq PF(MS) 15a assesses a participant's abilities and limitations with respect to everyday physical activities. Results are reported as a T-score. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 10 to 65. Higher T-scores represent higher physical function. Change from baseline in PROMIS PF score was analyzed using Mixed Effect Model for Repeated Measures (MMRM) to evaluate the result of the 2 periods (DBTP and DBE).
Time Frame: Baseline, Week 48, Week 96, Week 120, Week 144 and Week 156 (combined DBTP and DBE periods)
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure. The result reported for this outcome measure are the results from data of combined DBTP and DBE periods.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 551 | 545
units on a scale
  Week 48 | -0.30 [-0.79 to 0.19] | 0.05 [-0.45 to 0.55]
  Week 96 | -0.76 [-1.35 to -0.16] | -0.14 [-0.74 to 0.46]
  Week 120 | -0.29 [-0.95 to 0.37] | -0.25 [-0.92 to 0.42]
  Week 144 | -1.04 [-1.82 to -0.25] | -0.70 [-1.53 to 0.14]
  Week 156 | -1.61 [-2.70 to -0.51] | -1.44 [-2.66 to -0.23]

7. Secondary Outcome: DBTP and DBE Period: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Score at Week 48, Week 96, Week 120, Week 144 and Week 156
Description: PROMIS Fatigue score was assessed with PROMIS Short Form v1.0 - Fatigue - Multiple Sclerosis 8a (PROMIS Fatigue (MS) 8a). PROMIS Fatigue (MS) 8a assesses level of fatigue and its interference on daily activities. Results are reported as a T-score. In the general population, T-scores have a mean of 50, standard deviation of 10, and range from 33 to 85. Higher T-scores represent higher fatigue. Change from baseline in PROMIS fatigue score was analyzed using Mixed Effect Model for Repeated Measures (MMRM) to evaluate the result of the 2 periods (DBTP and DBE).
Time Frame: Baseline, Week 48, Week 96, Week 120, Week 144 and Week 156 (combined DBTP and DBE periods)
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 551 | 545
units on a scale
  Week 48 | -1.39 [-1.98 to -0.81] | -1.82 [-2.41 to -1.23]
  Week 96 | -1.60 [-2.32 to -0.87] | -2.14 [-2.88 to -1.41]
  Week 120 | -1.44 [-2.25 to -0.63] | -1.32 [-2.15 to -0.50]
  Week 144 | -1.88 [-2.90 to -0.86] | -0.98 [-2.06 to 0.10]
  Week 156 | 0.72 [-0.78 to 2.22] | -0.21 [-1.90 to 1.48]

8. Secondary Outcome: DBTP and DBE Period: Total Number of T1 Gadolinium-positive (Gd+) Lesions
Description: Analysis of Gadolinium-positive T1 lesions was done using magnetic resonance imaging (MRI) scans.
Time Frame: From baseline to 176 weeks
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Measure: Mean (95% Confidence Interval); unit: lesions per scan
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 564 | 560
lesions per scan | 0.35 [0.29 to 0.42] | 0.52 [0.43 to 0.62]

9. Secondary Outcome: DBTP and DBE Period: New or Enlarging T2 Lesions Rate
Description: Analysis of new or enlarging T2 lesions rate was done using magnetic resonance imaging (MRI) scans. Negative binomial model for lesion count (summed over scans) includes treatment and covariates based on randomization strata and baseline volume of T2 lesion (continuous), with offset equal to the log of the time in years between the last available MRI scan and the baseline scan.
Time Frame: From baseline to 176 weeks
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Measure: Mean (95% Confidence Interval); unit: lesions per year
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 564 | 560
lesions per year | 5.78 [5.02 to 6.65] | 5.45 [4.73 to 6.28]

10. Secondary Outcome: DBTP Period: Neurofilament Light Chain Concentration (NfL) at Week 12
Description: NfL is a biomarker of neuro-axonal damage whose concentration was assessed in blood at Week 12.
Time Frame: Week 12
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per liter (ng/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 533 | 528
nanogram per liter (ng/L) | 12.90 [12.48 to 13.34] | 12.88 [12.46 to 13.31]

11. Secondary Outcome: DBTP and DBE Periods: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Adverse Events of Special Interest (AESIs)
Description: Adverse event (AE): Any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the study drug. Serious AE: an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs: those AEs with an onset date on or after the date of first study intervention administration, or AEs present prior to any study intervention administration but exacerbating after. TEAEs included both Serious TEAEs and non-serious TEAEs. AESIs included liver AEs (possible drug-induced, non-infectious, non-alcoholic, and immune-mediated), infections (serious and opportunistic infections), lipase and amylase elevation, and seizure.
Time Frame: From baseline to 176 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 563 | 559
Participants
  Participants with TEAEs | 485 | 482
  Participants with AESIs | 120 | 117

12. Secondary Outcome: DBTP and DBE Periods: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: Severity of adverse events (AE) were assessed by the investigator per the National Cancer Institute- Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0. Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death. Number of participants with Grades 1, 2, 3, 4 and 5 were reported.
Time Frame: From baseline to 176 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 485 | 482
Participants
  Participants with Grade 1 | 50 | 56
  Participants with Grade 2 | 349 | 327
  Participants with Grade 3 | 82 | 88
  Participants with Grade 4 | 3 | 10
  Participants with Grade 5 | 1 | 1

13. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Diastolic Blood Pressure and Systolic Blood Pressure
Description: Diastolic blood pressure and systolic blood pressure were measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: diastolic blood pressure and systolic blood pressure from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 442 | 444
millimeter of mercury (mmHg)
  Systolic Blood Pressure | 2.6 (11.18) | 0.2 (10.83)
  Diastolic Blood Pressure | 1.8 (8.35) | 0.0 (8.67)

14. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: pulse rate from baseline up to baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 442 | 443
beats per minute | 2.6 (10.22) | 1.9 (9.68)

15. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Respiratory Rate
Description: Respiratory rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: respiratory rate from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 441 | 442
breaths per minute | -0.1 (1.76) | -0.2 (1.88)

16. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Weight
Description: Changes in vital signs: weight from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 442 | 443
kilograms (kg) | -0.21 (5.867) | 0.48 (5.490)

17. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Vital Signs: Temperature
Description: Temperature was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in vital signs: Temperature from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 443 | 442
degree Celsius | 0.00 (0.326) | 0.02 (0.319)

18. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Electrocardiograms (ECGs) Parameter: Heart Rate
Description: Heart rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in ECG parameter: heart rate from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 65 | 50
beats per minute | 3.0 (10.90) | -0.1 (12.55)

19. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Electrocardiograms (ECGs) Parameters: QT Interval - Fridericia's Correction Formula, PR Interval and QRS Duration
Description: QT Interval - Fridericia's Correction Formula, PR Interval and QRS Duration was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Changes in ECG parameter: QT Interval - Fridericia's Correction Formula, PR Interval and QRS Duration from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 65 | 50
milliseconds (msec)
  QT Interval - Fridericia's Correction Formula: number analyzed (Participants) | 65 | 49
  QT Interval - Fridericia's Correction Formula | -2.77 (16.005) | -1.37 (12.053)
  PR Interval | -5.2 (14.31) | -2.5 (14.65)
  QRS Duration | -3.7 (7.48) | -1.5 (10.82)

20. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Hemoglobin and Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: erythrocytes mean corpuscular HGB concentration and hemoglobin. Changes in hematology parameters: erythrocytes mean corpuscular HGB concentration and hemoglobin from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment. Here, Overall number of participants analyzed signifies those participants who were evaluable for this outcome measure and "number analyzed"= participants who were evaluable for the specified categories.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 433 | 432
gram per liter (g/L)
  Hemoglobin | -3.5 (10.74) | -2.8 (11.34)
  Erythrocytes Mean Corpuscular HGB Concentration: number analyzed (Participants) | 422 | 416
  Erythrocytes Mean Corpuscular HGB Concentration | -2.7 (12.43) | -1.0 (11.96)

21. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes and Reticulocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes and Reticulocytes. Changes in hematology parameters: Platelets, Leukocytes, Neutrophils, Eosinophils, Basophils, Monocytes, Lymphocytes and Reticulocytes from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 433 | 430
10^9 cells per liter
  Platelets: number analyzed (Participants) | 428 | 428
  Platelets | -4.8 (47.09) | 8.8 (53.83)
  Leukocytes | -0.17 (2.165) | -0.09 (1.958)
  Neutrophils: number analyzed (Participants) | 358 | 353
  Neutrophils | -0.316 (1.8846) | -0.210 (1.8356)
  Eosinophils: number analyzed (Participants) | 424 | 424
  Eosinophils | 0.0510 (0.15999) | 0.0203 (0.15853)
  Basophils: number analyzed (Participants) | 424 | 424
  Basophils | -0.0009 (0.03657) | -0.0003 (0.03786)
  Monocytes: number analyzed (Participants) | 424 | 424
  Monocytes | 0.0785 (0.18171) | 0.0656 (0.17816)
  Lymphocytes: number analyzed (Participants) | 424 | 424
  Lymphocytes | -0.0307 (0.58566) | -0.0401 (0.58108)
  Reticulocytes: number analyzed (Participants) | 411 | 411
  Reticulocytes | 0.488 (20.2014) | -0.827 (17.6824)

22. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Hematocrit. Changes in hematology parameter: Hematocrit from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 426 | 419
percentage of cells | -0.0069 (0.03359) | -0.0076 (0.03238)

23. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin. Changes in hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: picogram (pg)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 429 | 429
picogram (pg) | -0.61 (1.588) | -0.62 (1.956)

24. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume. Changes in hematology parameter: Erythrocytes Mean Corpuscular Volume from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 422 | 417
femtoliters | -1.42 (5.999) | -1.75 (4.895)

25. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Bilirubin and Creatinine
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Bilirubin and Creatinine. Changes in biochemistry parameters: Bilirubin and Creatinine from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 435 | 439
micromoles per liter (mcmol/L)
  Bilirubin: number analyzed (Participants) | 433 | 439
  Bilirubin | -0.08 (4.792) | 0.15 (4.792)
  Creatinine: number analyzed (Participants) | 435 | 438
  Creatinine | 0.6 (12.76) | 2.4 (8.67)

26. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase. Changes in biochemistry parameters: Aspartate Aminotransferase, Alanine Aminotransferase, Alkaline Phosphatase, Amylase, Lipase, Gamma Glutamyl Transferase and Lactate Dehydrogenase from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 435 | 440
units per liter (U/L)
  Aspartate Aminotransferase: number analyzed (Participants) | 433 | 433
  Aspartate Aminotransferase | 2.32 (18.190) | 6.49 (64.249)
  Alanine Aminotransferase: number analyzed (Participants) | 433 | 438
  Alanine Aminotransferase | 4.06 (23.308) | 8.55 (52.866)
  Alkaline Phosphatase | 4.20 (23.289) | 7.65 (20.252)
  Amylase: number analyzed (Participants) | 434 | 439
  Amylase | -0.5 (17.04) | 2.8 (16.84)
  Lipase: number analyzed (Participants) | 435 | 438
  Lipase | -2.5 (33.36) | 3.5 (17.33)
  Gamma Glutamyl Transferase: number analyzed (Participants) | 375 | 390
  Gamma Glutamyl Transferase | 4.28 (21.091) | 5.51 (40.098)
  Lactate Dehydrogenase: number analyzed (Participants) | 431 | 430
  Lactate Dehydrogenase | 6.16 (28.235) | -4.53 (26.014)

27. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Sodium, Potassium, Calcium, Magnesium, Glucose, Chloride, Urea Nitrogen, Phosphate, Bicarbonate and Corrected Calcium
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Sodium, Potassium, Calcium, Magnesium, Glucose, Chloride, Urea Nitrogen, Phosphate, Bicarbonate and Corrected Calcium. Changes in biochemistry parameters: Sodium, Potassium, Calcium, Magnesium, Glucose, Chloride, Urea Nitrogen, Phosphate, Bicarbonate and Corrected Calcium from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 436 | 439
millimole per liter (mmol/L)
  Sodium | 0.9128 (2.34334) | 0.7904 (2.28990)
  Potassium: number analyzed (Participants) | 436 | 438
  Potassium | 0.0320 (0.43741) | 0.0893 (0.42341)
  Calcium: number analyzed (Participants) | 435 | 438
  Calcium | 0.004 (0.1139) | -0.002 (0.1029)
  Magnesium: number analyzed (Participants) | 435 | 438
  Magnesium | 0.004 (0.0682) | 0.002 (0.0656)
  Glucose: number analyzed (Participants) | 432 | 437
  Glucose | 0.06 (0.928) | 0.25 (1.146)
  Chloride: number analyzed (Participants) | 435 | 438
  Chloride | 1.8 (3.42) | 1.7 (2.95)
  Urea Nitrogen: number analyzed (Participants) | 434 | 437
  Urea Nitrogen | 0.222 (1.2668) | 0.114 (1.2654)
  Phosphate: number analyzed (Participants) | 432 | 435
  Phosphate | -0.053 (0.2048) | -0.026 (0.1724)
  Bicarbonate: number analyzed (Participants) | 359 | 375
  Bicarbonate | 0.05 (2.561) | 0.04 (2.725)
  Corrected Calcium: number analyzed (Participants) | 434 | 437
  Corrected Calcium | 0.0297 (0.09428) | 0.0317 (0.09071)

28. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameters: Total Protein and Albumin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameters: Total Protein and Albumin. Changes in biochemistry parameters: Total Protein and Albumin from baseline up to 176 weeks were reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 436 | 439
gram per liter (g/L)
  Total protein: number analyzed (Participants) | 432 | 438
  Total protein | -1.26 (4.865) | -0.47 (4.417)
  Albumin | -1.28 (3.520) | -1.67 (3.284)

29. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Biochemistry Parameter: Glomerular Filtration Rate
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the biochemistry parameter: Glomerular Filtration Rate. Changes in biochemistry parameter: Glomerular Filtration Rate from baseline up to 176 weeks was reported. The Glomerular Filtration Rate will be measured as milliliter per minute per 1.73 square meter (mL/min/1.73m^2).
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 376 | 374
mL/min/1.73m^2 | -3.3 (13.82) | -5.6 (13.54)

30. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Urinalyses Parameter: Potential of Hydrogen (pH) of Urine
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameter: pH. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 - 6.0). Changes in urinalyses parameter: pH from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 428 | 436
pH | -0.08 (0.886) | 0.01 (0.913)

31. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Urinalyses Parameter: Specific Gravity of Urine
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameter: Specific Gravity of Urine. Changes in urinalyses parameter: Specific Gravity of Urine from baseline up to 176 weeks was reported.
Time Frame: From baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Kilogram per cubic meter
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 429 | 436
Kilogram per cubic meter | 0.0006 (0.03891) | 0.0011 (0.02189)

32. Secondary Outcome: DBTP and DBE Periods: Absolute Concentrations of Immunoglobulin (Ig) Levels
Description: Absolute Concentrations serum levels of IgG, IgA, IgM were assessed.
Time Frame: At Week 176
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 360 | 366
gram per liter (g/L)
  IgA | 1.750 (0.7987) | 2.503 (1.0582)
  IgG | 9.693 (2.1096) | 10.529 (2.2363)
  IgM | 1.101 (0.6096) | 1.181 (0.6619)

33. Secondary Outcome: DBTP and DBE Periods: Change From Baseline in Immunoglobulin (Ig) Levels
Description: Change from baseline serum levels of IgG, IgA, IgM were assessed.
Time Frame: Baseline to 176 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Teriflunomide | Evobrutinib
Number analyzed (Participants) | 355 | 362
gram per liter (g/L)
  IgA | -0.262 (0.3572) | 0.483 (0.5320)
  IgG | -0.733 (1.4414) | 0.105 (1.4556)
  IgM | -0.165 (0.2979) | -0.187 (0.2794)

34. Secondary Outcome: OLE Period: Annualized Relapse Rate (ARR)
Description: The qualifying relapse is the occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis (MS) (for more than [>] 24 hours, no fever, infection, injury, AEs, and preceded by a stable or improving neurological state for more than or equal to [>=] 30 days).
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment.
Measure: Mean (95% Confidence Interval); unit: relapses per year
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
relapses per year | NA [NA to NA] — NA signifies data is not available as no participant in this arm group had a relapse.

35. Secondary Outcome: OLE Period: Percentage of Participants Without 24-Week Confirmed Disability Progression (CDP) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability progression was defined as increase in EDSS of greater than or equal to [>=] 1 point from baseline EDSS score, if EDSS score at baseline is 5.0 or less and an increase of >=0.5 point, if the baseline score is 5.5. Disability progression is considered sustained for 24 weeks when the initial increase in the EDSS is confirmed at a regularly scheduled visit at least 24 weeks after the initial documentation of neurological worsening. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis).
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. No participants with confirmed disability progression sustained for 24 weeks as measured on EDSS.
Measure: Number; unit: percentage of participants
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
percentage of participants | 0

36. Secondary Outcome: OLE Period: Percentage of Participants With 24-Week Confirmed Disability Improvement (CDI) as Measured by Expanded Disability Status Scale (EDSS)
Description: Disability improvement was defined as a reduction of 1 point from Baseline EDSS score when the Baseline score is >= 2 and less than or equal to [<=] 6 and a reduction of 0.5 point from Baseline EDSS score when the Baseline score is >= 6.5 and <= 9.5. Disability improvement is considered sustained when the initial reduction in the EDSS score is confirmed at a regularly scheduled visit at least 24 weeks after the initial reduction. The total EDSS score ranges from 0 (normal) to 10 (death due to multiple sclerosis).
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: Full analysis Set (FAS) included all participants who were randomized to study treatment. No participants did not meet the baseline criteria of EDSS >=2.
Measure: Number; unit: percentage of participants
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
percentage of participants | 0

37. Secondary Outcome: OLE Period: Symbol Digit Modalities Test (SDMT)
Description: The SDMT is a test of information processing speed. It consists of 9 abstract symbols. Each symbol is paired with a single digit. The participant is provided with a "key", showing each symbol digit pair. In addition, the participants are shown several rows of the 9 symbols, which are arranged pseudo-randomly, without the digit. Participants are asked to voice the digit associated with each symbol as rapidly as possible for 90 seconds. The SDMT score ranges from 0 to 110 where higher scores indicated improvement and lower scores indicated worsening. Participant wise data was reported for this outcome measure.
Time Frame: Assessed from OLE baseline to OLE Week 96; OLE Week 48 were reported for Participants 1 and 2 and OLE Week 12 were reported for Participant 3
Population: Full Analysis Set (FAS) included all participants who were randomized to study treatment. No summary analysis was done as study was prematurely terminated and participant wise data was reported. Here, "number analyzed" signifies specific participant evaluated in the arm of this outcome measure.
Measure: Number; unit: units on a scale
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
units on a scale
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 60
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 40
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 50

38. Secondary Outcome: OLE Period: Change From Baseline in PROMISnq Physical Function (PF) Multiple Sclerosis (MS) 15a at Week 52
Description: Physical function was assessed with PROMISnq Short Form v2.0 - Physical Function - Multiple Sclerosis 15a (PROMISnq PF(MS) 15a). PROMISnq PF(MS) 15a assesses a participant's abilities and limitations with respect to everyday physical activities. Results are reported as a T-score. In the general population, T-scores have a mean of 50, standard deviation of 10, and ranges from 10 to 65. Higher T-scores represent higher physical function. Participant wise data was reported for this outcome measure.
Time Frame: OLE Baseline (DBTP Week 96), OLE Week 52
Population: as for outcome 37
Measure: Number; unit: T-score
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
T-score
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 52
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 63
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 51

39. Secondary Outcome: OLE Period: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue (MS) 8a Score at Week 52
Description: PROMIS Fatigue score was assessed with PROMIS Short Form v1.0 - Fatigue - Multiple Sclerosis 8a (PROMIS Fatigue (MS) 8a). PROMIS Fatigue (MS) 8a assesses level of fatigue and its interference on daily activities. Results are reported as a T-score. In general, T-scores have a mean of 50, standard deviation of 10, and range from 33 to 85. Higher T-scores represent higher fatigue. Participant wise data was reported for this outcome measure.
Time Frame: OLE baseline (DBTP Week 96), OLE Week 52
Population: as for outcome 37
Measure: Number; unit: T-score
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
T-score
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 43
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 42
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 41

40. Secondary Outcome: OLE Period: Number of Participants With Abnormalities in Laboratory Parameters
Description: Laboratory investigation included hematology, biochemistry and coagulation. The number of participants with abnormalities in laboratory parameters were reported.
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
Participants
  Hematology | 1
  Biochemistry | 1
  Coagulation | 0

41. Secondary Outcome: OLE Period: Number of Participants With Abnormalities in Vital Signs
Description: Vital signs included temperature, pulse rate, respiration rate and blood pressure and weight (taken after 5 minutes in the sitting position). The number of participants with abnormalities in vital signs were reported.
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
Participants | 0

42. Secondary Outcome: OLE Period: Number of Participants With Abnormalities in Electrocardiograms (ECGs) Findings
Description: ECG recordings included, heart rate, PR interval and QRS duration. ECG recordings were obtained after the participants have rested for at least 5 minutes in supine position. The number of participants with abnormalities in ECG findings were reported.
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
Participants | 1

43. Secondary Outcome: OLE Period: Number of New or Enlarging T2 Lesions
Description: Analysis of number of new or enlarging T2 lesions was done using magnetic resonance imaging (MRI) scans. Negative binomial model for lesion count (summed over scans) includes treatment and covariates based on randomization strata and baseline volume of T2 lesion (continuous), with offset equal to the log of the time in years between the last available MRI scan and the baseline scan. Participant wise data was reported for this outcome measure.
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: as for outcome 37
Measure: Number; unit: number of lesions
Units Other Than Participants: lesions
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
Number analyzed (lesions) | 33
number of lesions
  Participant 1: number analyzed (Participants) | 1
  Participant 1: number analyzed (lesions) | 11
  Participant 1 | 11
  Participant 2: number analyzed (Participants) | 1
  Participant 2: number analyzed (lesions) | 11
  Participant 2 | 0
  Participant 3: number analyzed (Participants) | 1
  Participant 3: number analyzed (lesions) | 11
  Participant 3 | 0

44. Secondary Outcome: OLE Period: Change From Baseline in T2 Lesion Volume
Description: Change from baseline in T2 lesion volume was reported. Participant wise data was reported for this outcome measure.
Time Frame: From OLE baseline (DBTP Week 96) to OLE Week 52
Population: as for outcome 37
Measure: Number; unit: milliliter (mL)
Arm/Group | Evobrutinib
Number analyzed (Participants) | 3
milliliter (mL)
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 0.471
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | -0.111
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 0

ADVERSE EVENTS:
Time Frame: From baseline to 176 weeks
Description: Safety (SAF) analysis set included all participants who received at least one dose of study treatment.
Arm/Group | Teriflunomide | Evobrutinib
All-Cause Mortality (participants affected / at risk) | 1/563 | 1/559
Serious Adverse Events (participants affected / at risk) | 33/563 | 45/559
Other Adverse Events (participants affected / at risk) | 409/563 | 361/559
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide (N=563) | Evobrutinib (N=559)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 1 (1)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Blast injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Impacted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 3 (3) | 4 (4)
Neurologic neglect syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Abortion complete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Psychogenic movement disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriflunomide (N=563) | Evobrutinib (N=559)
Leukopenia (Blood and lymphatic system disorders) | 39 (66) | 13 (15)
Neutropenia (Blood and lymphatic system disorders) | 41 (87) | 20 (23)
Diarrhoea (Gastrointestinal disorders) | 53 (71) | 15 (20)
Fatigue (General disorders) | 32 (34) | 29 (33)
COVID-19 (Infections and infestations) | 108 (117) | 121 (142)
Nasopharyngitis (Infections and infestations) | 61 (82) | 67 (105)
Upper respiratory tract infection (Infections and infestations) | 42 (62) | 36 (56)
Urinary tract infection (Infections and infestations) | 26 (32) | 36 (56)
Alanine aminotransferase increased (Investigations) | 86 (134) | 77 (131)
Aspartate aminotransferase increased (Investigations) | 54 (71) | 51 (66)
Lipase increased (Investigations) | 35 (50) | 23 (31)
Neutrophil count decreased (Investigations) | 50 (83) | 25 (34)
White blood cell count decreased (Investigations) | 29 (38) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (28) | 34 (46)
Headache (Nervous system disorders) | 75 (175) | 81 (151)
Alopecia (Skin and subcutaneous tissue disorders) | 59 (63) | 32 (34)
Hypertension (Vascular disorders) | 32 (40) | 15 (19)

LIMITATIONS AND CAVEATS:
The Final Analysis represents the analysis of the cumulative data collected up to the Primary Analysis trigger and beyond through DBE up to the final database lock. Therefore, the endpoints were evaluated considering a time period from the start of DBTP to the end of the DBE Period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT04338022/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT04338022/SAP_001.pdf